CLINICAL TRIAL: NCT03652844
Title: A Multi-Phase, Prospective, Multi-Center, Single-Blind, Clinical Study to Evaluate the Safety and Efficacy of Allograft Adipose Matrix (AAM) and Diluted AAM for Pre-Jowl and Malar Augmentation to Correct Age Related Volume Deficit in the Face
Brief Title: Use of AAM for Correction of Age Related Volume Deficits in the Face
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Musculoskeletal Transplant Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MTF 18-04-01
Record Dates: First submitted 2018-08-28; First posted 2018-08-29 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Age-Related Atrophy

STUDY DESIGN:
Intervention Model Description: Randomized cohorts
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Allograft Adipose Matrix (AAM) 1.0 (Active Comparator)
  Interventions: Procedure: AAM
- Allograft Adipose Matrix (AAM) Diluted (Active Comparator)
  Interventions: Procedure: AAM

INTERVENTIONS:
Procedure: AAM — Subcutaneous injection procedure

SUMMARY:
The purpose of this study is to evaluate Allograft Adipose Matrix (AAM) in the face of people with age-related volume deficit - fat loss. AAM is a tissue used to correct fat loss. Participation in this study requires injections for placing AAM in the bilateral pre-jowl and malar areas of the face. The research will tell whether AAM is effective in maintaining mid-face fullness and whether the appearance of the skin improves after injection.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women, 30-70 years of age
2. Has overall mid-facial volume deficit of Grade 3 or 4 on Medicis Midface Volume Scale (MMVS)
3. Willingness and ability to provide written informed consent
4. Has not had AAM injected above the neck
5. Ability to understand and comply with the requirements of the study
6. Negative urine pregnancy test results at the time of study entry (if applicable).
7. Willingness to stay on consistent and current skin care regimen for the duration of the study
8. Willingness to maintain consistent and current diet and exercise for the duration of the study
9. Willingness to forego any cosmetic augmentation procedure for the duration of the study
10. Willingness to be photographed for educational, medical publication and other non-commercial purposes
11. Has BMI ≥18 and ≤30

Exclusion Criteria:

1. A subject with any uncontrolled systemic disease.
2. A subject in whom therapy for a systemic disease is not yet stabilized will not be considered for entry into the study.
3. A subject with a significant history or current evidence of a medical, psychological or other disorder that, in the investigator's opinion, would preclude enrollment into the study.
4. Women that are pregnant, nursing, or planning a pregnancy during the duration of the study
5. A subject that has had AAM injected above the neck
6. A subject unwilling to be photographed for educational, medical publication and other non-commercial purposes
7. A subject with a history of diabetes
8. A subject with known hypersensitivity to any of the components of AAM
9. A subject that has had, or who knowingly will have, dental work +/- 4 weeks prior to, or following AAM injection
10. A subject using any systemic corticosteroid or immunosuppressive medications within 30 days prior to treatment and topical steroids on the face within 14 days prior to treatment and throughout the study
11. A subject that has participated in another research study within 30 days of enrollment in this study
12. A subject that is unwilling to forego any cosmetic augmentation treatment for the duration of the study
13. A subject that has been treated with Botulinum Toxin below the orbital rim within 6 months of study entry.
14. A subject that is unwilling to forego cosmetic facial treatments for the duration of the study
15. A subject that has received Sculptra in the treatment area
16. A subject that has received dermal filler in the treatment area within 2 years prior to randomization
17. A subject that has previously undergone mid-face cosmetic plastic surgery, tissue grafting, or tissue augmentation with silicone, semi-permanent fillers or fat
18. A subject that has previously undergone laser resurfacing, intense pulsed light treatment, chemical peel, or other ablative or non-ablative treatment within 6 months
19. Subject is immunocompromised or immunosuppressed
20. History of keloid formation or hypertrophic scars
21. NSAID or Aspirin, other than a stable low dose aspirin regimen, within 1 week (7 days) prior to treatment
22. Concomitant anticoagulant therapy, antiplatelet therapy, or history of bleeding disorders or connective tissue disorders
23. A subject with recent excessive facial exposure to sunlight or artificial UV light (e.g.: use of tanning beds/booths and/or sunbathing)
24. A subject with a recent history or active presence of any facial skin condition/disease that might interfere with the diagnosis or evaluation of study parameters (i.e. moderate to severe acne vulgaris, atopic dermatitis, psoriasis, rosacea, seborrheic dermatitis, excessive facial hair or coloration)
25. Current participation or participation within 30 days prior to the start of this study in a drug or other investigational research study
26. A subject not deemed to be enrolled at the discretion of the surgeon investigator

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-08-27 (Actual); Primary Completion 2019-07-12 (Actual); Study Completion 2019-07-12 (Actual)

PRIMARY OUTCOMES:
Volume change for the treated areas using the validated 4 point MEDICIS Mid-Face Volume Scale Assessment (MMVSA) at 24 weeks post-treatment compared to pre-treatment | 24 weeks
  MMVSA measures facial volume deficit, ranging from 1 (fairly full midface) to 4 (substantial loss of fullness in the midface area). Lower values represent a better outcome.
Three-D facial photography (Canfield) with computation of volume changes at 24 weeks compared to pre-treatment. | 24 weeks

SECONDARY OUTCOMES:
Duration of effectiveness when the average of the Evaluating Investigators' live assessments of the MMVSA scale will return to, or be worse than, the pre-treatment level over 24 weeks post-treatment. | 24 weeks
  MMVSA measures facial volume deficit, ranging from 1 (fairly full midface) to 4 (substantial loss of fullness in the midface area). Lower values represent a better outcome.
Volume change assessments using the Global Aesthetic Improvement Scale (GAIS) at 24 weeks post-treatment compared to pre-treatment | 24 weeks
  GAIS rates improvement in appearance. Scores range from 0 (worse) to 4 (very much improved). Higher values represent a better outcome.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Aesthetic Eyelid Plastic Surgery, Boca Raton, Florida
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - Dallas Plastic Surgery Institute, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No